CLINICAL TRIAL: NCT05218863
Title: Incidence, Diagnosis, Management and Outcome of Acute Mesenteric Ischaemia: a Prospective, Multicentre Observational Study
Brief Title: Incidence, Diagnosis, Management and Outcome of Acute Mesenteric Ischemia
Acronym: AMESI
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Annika Reintam Blaser, A/Professor, University of Tartu
Other Study IDs: AMESI Study
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Acute Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed AMI: Patients in whom diagnosis of acute mesenteric ischaemia (AMI) was confirmed. For these patients full data collection is required, including 1-year outcome. Maximum 500 patients in this group.
  Interventions: Other: No intervention
- AMI suspected but not confirmed: Patients in whom acute mesenteric ischaemia (AMI) was suspected but not confirmed. For these patients minimal data will be collected, only hospital survival as outcome.
  Maximum 2000 patients in this group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a prospective, multicentre observational study screening all adult patients admitted to a participating hospital over a 6-month study period (may be adjusted to 4-8 months according to recruitment) and including all patients with suspicion of or confirmed acute mesenteric ischaemia (AMI).

Only admission data and hospital mortality outcome will be collected for patients in whom suspicion of AMI is not confirmed. For patients with confirmed AMI full data collection regarding diagnostics, management and long-term outcome is required.

Investigators aim to recruit 40-50 sites with expected median of 10-20 patients with confirmed AMI per site during the study period (naturally depending on the size of the hospital). The start of the study is planned for Spring 2022.

The aim of the study is to identify the incidence of AMI and its different forms in adult hospitalized patients, and to describe patient characteristics (demographic, clinical and laboratory) at baseline, applied diagnostics and management, as well as outcomes in patients with AMI. An additional aim is to compare the baseline characteristics and outcomes of patients with confirmed AMI to those of patients with suspected AMI in whom the diagnosis was not confirmed.

ELIGIBILITY:
Inclusion Criteria:

All patients with suspected AMI

Exclusion Criteria:

Age <18 years Consent declined by patient or next of kin Chronic mesenteric ischaemia without an acute event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to a participating hospital during the study period will be screened to include all patients with suspicion of or confirmed acute mesenteric ischaemia (AMI).
  All patients with suspicion of or confirmed AMI are to be included in the study in accordance with local ethics requirements:
  * If suspicion of AMI is NOT confirmed, only baseline data and hospital mortality outcome is collected
  * if the diagnosis of AMI is confirmed, then full data collection is required
Sampling Method: Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of AMI | 6 months
  Incidence of AMI in hospitalized adult patients in acute care hospitals

SECONDARY OUTCOMES:
30 days survival of AMI | 30 days after admission/suspicion of AMI/study inclusion
  survival of patients with confirmed AMI
Proportion of different forms of AMI | 6 months
  Proportion of each form of AMI from all AMI cases
Time to diagnosis | through study completion, study duration 6 months
  Time from symptoms to diagnosis
Time to treatment | through study completion, study duration 6 months
  Time from diagnosis to treatment
Treatment | through study completion, study duration 6 months
  Surgery, endovascular intervention or palliation
1 year survival | 1 year
  Survival of patients with AMI 1 year after diagnosis
Quality of life score | 1 year
  EQ-5D-5L (EuroQoL - European Quality of Life ), 5-25 points, the lower score means better outcome

CONTACTS AND LOCATIONS:
Locations (3):
- Estonia (2):
  - North Estonian Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Kantonsspital Luzern, Lucerne, Switzerland

REFERENCES:
- [Derived] Acosta S, Blaser AR, Nuzzo A, Soltanzadeh-Naderi Y, Starkopf J, Forbes A, Murruste M, Tamme K, Voomets AL, Koitmae M, Bala M, Bodnar Z, Casian D, Demetrashvili Z, Biloslavo A, Munoz-Cruzado VD, Hess B, Kase K, Kirov M, Lindner M, Loudet CI, Damaskos D, Bjorck M; AMESI Investigators (Collaborators). D-Dimer in Acute Mesenteric Venous Thrombosis: A Prospective Case-Control International Multicenter Study. Biomark Insights. 2024 Nov 26;19:11772719241296631. doi: 10.1177/11772719241296631. eCollection 2024. PMID 39600492
- [Derived] Reintam Blaser A, Mandul M, Bjorck M, Acosta S, Bala M, Bodnar Z, Casian D, Demetrashvili Z, D'Oria M, Duran Munoz-Cruzado V, Forbes A, Fuglseth H, Hellerman Itzhaki M, Hess B, Kase K, Kirov M, Lein K, Lindner M, Loudet CI, Mole DJ, Murruste M, Nuzzo A, Saar S, Scheiterle M, Starkopf J, Talving P, Voomets AL, Voon KKT, Yunus MA, Tamme K; AMESI Investigators (Collaborators). Incidence, diagnosis, management and outcome of acute mesenteric ischaemia: a prospective, multicentre observational study (AMESI Study). Crit Care. 2024 Jan 23;28(1):32. doi: 10.1186/s13054-024-04807-4. PMID 38263058